CLINICAL TRIAL: NCT04073524
Title: The Wild Man Programme. A Nature-based Rehabilitation Enhancing Quality of Life for Men on Long-term Sick Leave - a Matched Controlled Study
Brief Title: The Wild Man Programme - a Nature-based Rehabilitation Enhancing Quality of Life for Men on Long-term Sick Leave
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Southern Denmark (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: USouthernDenmarkpsychology
Record Dates: First submitted 2019-08-23; First posted 2019-08-29 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Stress; Anxiety; Depression; Cardiac Disease; Cancer; Diabetes; Copd
Keywords: Supportive Environment Theory (SET); Aesthetic Affective Theory (AAT); Attention Restoration Theory (ART); Nature-Body-Mind-Community (NBMC)
MeSH Terms: conditions — Anxiety Disorders; Depression; Heart Diseases; Neoplasms; Diabetes Mellitus; Pulmonary Disease, Chronic Obstructive | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The study is a matched control study where the intervention group receives a nine-week nature-based intervention and is compared to a matched control group receiving case management as treatment as usual in the municipalities (see figure 1). All primary and secondary outcomes are measured at baseline (T1), post treatment (T2), and at follow-up 6 months post intervention (T3).
Masking Description: The municipality of Svendborg has the superior responsibility for the 'Wild man programme'. Participation in the intervention as well as participation in the study is voluntary. All information collected in the study will be treated confidentially, and participation requires a signed consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature-Body-Mind-Community (NBMC) + treatment as usual (Experimental): 9 weeks of nature-based therapy (Nature-Body-Mind-Community (NBMC)) treatment as usual
  Interventions: Other: Nature-Body-Mind-Community; Other: Treatment as usual
- Treatment as usual (Other): Treatment as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Nature-Body-Mind-Community — The Nature-Body-Mind-Community (NBMC) approach has been developed in a pilot project over 2014-2018. The 'Wild man Programme' consists of the following main elements: 1. Nature environments and nature experiences, 2. Mind relaxation and meditation, 3. Body awareness and 4. Fire talks, storytelling and community spirit.
  Arms: Nature-Body-Mind-Community (NBMC) + treatment as usual
Other: Treatment as usual — Treatment as usual consist of the rehabilitation offered by the hospital or municipality for the specific condition e.i. cancer, diabetes, COPD, anxiety, depression and stress

SUMMARY:
The aim of the present study is to examine whether the nature based 'Wild man Programme' can help to increase quality of life among men on sick leave compared to treatment as usual. Additionally, the study examines which natural environments best work as supportive environments in the rehabilitation.

DETAILED DESCRIPTION:
Many men in Denmark have poor mental health and need help to recover. However, designing a rehabilitation intervention appealing to men is challenging. The 'Wild man Programme' is a rehabilitation programme for men on long-term sick leave and with clinical or self-reported stress due to prolonged health problems such as stress, anxiety, depression, cancer, chronic obstructive pulmonary disease (COPD), cardiovascular disease or diabetes. The programme is a nature-based rehabilitation (NBR) initiative combining nature experiences, attention training, body awareness training and supporting community spirit.

The aim of the present study is to examine whether the 'Wild man Programme' can help to increase quality of life among men on sick leave compared to treatment as usual. Additionally, the study examines which natural environments best work as supportive environments in the rehabilitation.

A matched control study comparing an intervention group (N=38) which receives a nine-week nature-based intervention to a control group (N=38) receiving case management as treatment as usual in the municipalities. Outcomes are measured at baseline (T1), post treatment (T2), and at follow-up 6 months post intervention (T3). The primary outcome is an improvement in quality of life and the secondary outcome is a decrease in stress level.

With the 'Wild man Programme' we investigate whether it is a model that can be implemented in the health system in Denmark to help men with different kinds of health problems improve their quality of life and stress levels. The programme can also deliver valuable information for future nature-based rehabilitation for women (Wild woman) and mixed gender groups. The project will also contribute with information on whether the method and the concept can be a valuable tool for health professionals in the health sector.

ELIGIBILITY:
The inclusion and exclusion criteria are similar for the two groups.

The inclusion criteria are:

* male gender
* 18 to 68 years of age
* clinical or self-reported symptoms of stress, anxiety, depression
* clinical diagnosis of cancer, cardiovascular disease, chronic obstructive pulmonary disease (COPD), diabetes or other kinds of chronic diseases
* ability to walk approximately three kilometers in nature
* ability to understand and speak Danish

The exclusion criteria are:

- psychosis or psychotic disorders, brain injuries or physical disabilities that prevent the participant from participating in the physical exercise programme or move about in nature

Ages: 18 Years to 68 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Level of quality of life - total score | 9 weeks
  The primary outcome is self-experienced quality of life. The World Health Organization's brief quality of life questionnaire (WHOQOL-BREF) will be used. The questionnaire examines four domains on a five-point Likert scale: Physical health, mental health, social relationships and health-related environments e.g. instant access to medical care. The global quality of life is based on the participants' scores on the four domains and they range from 0-100, with a high score indicating high quality of life.

SECONDARY OUTCOMES:
Level of quality of life - physical health | 9 weeks
  The WHOQOL-BREF will be used. The domain of physical health is measured on a five-point Likert scale with five questions.
Level of quality of life - mental health | 9 weeks
  The WHOQOL-BREF will be used. The domain of mental health is measured on a five-point Likert scale with five questions.
Level of quality of life - social relationships | 9 weeks
  The WHOQOL-BREF will be used. The domain of social relationships is measured on a five-point Likert scale with five questions.
Level of quality of life - health related environments | 9 weeks
  The WHOQOL-BREF will be used. The domain of health related environments is measured on a five-point Likert scale with five questions.
Level of self-experienced restitution | 9 weeks
  Self-experienced restitution. The Perceived Restorativeness Scale-11 (PRS-11) will be used.
Level of self perceived stress | 9 weeks
  Self perceived stress. The Cohen's Perceived Stress Scale (PSS) will be used. The scale consists of 14 items measured on a five-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Høegmark, Master, Principal Investigator — University of Southern Denmark
Locations (1):
- Southern Danish University, Odense, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be submitted to the peer-reviewed journal BMC Public Health
Supporting Information: Study Protocol
Time Frame: The protocol paper will be submitted to BMC Public Health, June 2019. A a paper on the narratives of the participating men in the 'Wild man programme' will be submitted to Qualitative Health Research in June 2020. Finally, a paper on spontaneous attention in outdoor environments and change in quality of life will be submitted to Clinical Psychology in December 2020.
Access Criteria: Access to data is restricted due to the European laws. Please contact the Principal Investigator for more information.

REFERENCES:
- [Background] Bratland-Sanda, S., Andersson, E., Best, J., Høegmark, S. & Roessler, K. K. The use of physical activity, sport and outdoor life as tools of psychosocial intervention: the Nordic perspective 2019. Sport in Society. 22, 4, s. 654-670, 2018.